CLINICAL TRIAL: NCT02574494
Title: Does Breastfeeding Lower Blood Pressure in Postpartum Hypertensive Patients
Status: Completed | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Sarah Kilpatrick, Chair, Department of Obstetrics and Gynecology, Cedars-Sinai Medical Center
Other Study IDs: Pro00040747
Record Dates: First submitted 2015-10-04; First posted 2015-10-14 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Breastfeeding; Hypertension
MeSH Terms: conditions — Breast Feeding; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary aim is to establish whether breastfeeding is associated with lowering blood pressure in hypertensive women.

DETAILED DESCRIPTION:
Patients included in this study will have chosen to breastfeed.

1. The investigators will identify patients that are planning to breastfeed from their intake questionnaire that all patients receive upon admission to labor and delivery. They will also identify breastfeeding patients while performing our postpartum rounding.
2. The investigators will perform a chart review to determine their co-morbidities and current medications. Specifically, the patient information recorded will be age, parity, gestational age, delivery route, vital signs, medications, race, whether they are breastfeeding. Of note, all of the individuals listed to participate in this study have routine access to the patient's charts since they will be working with the patients regardless of their participation in the study.
3. Only hypertensive women will be included. Hypertension is defined as persistent Systolic blood pressure > 140 and or persistent diastolic blood pressure > 90.
4. Once it has been determined that they have met the inclusion criteria for the study the investigators will ask the patient's attending physician if we can approach the patient and explain the study and obtain consent.
5. Once consent is obtained, the investigators will inform the nurse. The patient will have her blood pressure taken prior to breastfeeding, during breastfeeding, and 1-2 hours after breastfeeding. This will occur 3 times in the postpartum period.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria include hypertensive women in the first 72 hours postpartum. The gestational age at delivery must be greater or equal to 34wk and the patient must be breastfeeding and/or pumping milk. The study will include patient's on anti-hypertensive. The study will also include patients receiving postpartum IV magnesium but they will have their blood pressure taken two times while on magnesium and two times after the magnesium has been discontinued.

Exclusion Criteria:

* The study will exclude patient's on dopamine agonist medications or HIV positive.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include breastfeeding mothers that have met criteria for hypertension.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-10; Primary Completion 2017-04 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Decrease in blood pressure after breastfeeding | Up to 16 months
  A decrease of 15mmHg systolic, 10mmHg diastolic, or a decrease of 10% from baseline will be considered significant.

OTHER OUTCOMES:
Blood pressure measurement | Up to 16 months
  Blood pressure will be measured using millimeters of mercury (mmHg).

CONTACTS AND LOCATIONS:
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States